CLINICAL TRIAL: NCT05630898
Title: Congenital Cytomegalovirus: Prevalence in Buenos Aires City
Brief Title: Congenital Cytomegalovirus: Prevalence in Buenos Aires City (cCMV Prevalence)
Acronym: cCMV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Daniela Satragno, MD, MD, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: HNinosBuenosAires
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Congenital Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva Swab for CMV PCR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMV PCR — Saliva CMV PCR

SUMMARY:
The goal of this observational study is to recognise the prevalnce of congenital cytomegalovirus (cCMV) and to follow up positive babies until 12 months The main questions it aims to answer are: pevalence of cCMV, cCMV clinicals outcomes during the first year of life.

Participants will be screened with a salive swab for CMV DNA. Babies with positive results will be follow up for one year.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is a frequent cause of congenital infection and a leading nongenetic cause of sensorineural hearing loss. In most infants with congenital CMV infection, clinical abnormalities do not manifest at birth; rather, the infection is asymptomatic. However, sensorineural hearing loss eventually develops in approximately 10 to 15% of CMV positive children.

The prevalence of congenital cytomegalovirus has been reported as 0·2% to 2·0% (average of 0·64%). There is not any publication of the prevalence of cCMV in Buenos Aires City. We aim the study to find the prevalence in this population Screening of newborns for CMV infection permit early identification of at-risk congenitally infected infants for purposes of targeted monitoring and intervention during critical stages of speech and language development.

Testing saliva via DNA detection of the virus through polymerase chain reaction testing (PCR) or rapid culture is shown to have a high sensitivity (>97%) and specificity (99%) for detecting congenital CMV infection.

Our objective is to describe the prevalence of cCMV using saliva specimens for PCR detection.

Secondary objectives includes describing prevalence of neurosensorial hearing loss and visual impairments during 1 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Newborns between 1 and 21 days
* informed consent

Exclusion Criteria:

* Lethal malformation

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of cCMV | 5 months
  newborns positive for CMV

SECONDARY OUTCOMES:
incidence of neurosensorial hearing loss during the 1° year of life | 1 year
  fail Hearing test
incidence of visual impairments detected during the 1° year of life | 1 year
  anormal eye exam

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Satragno, MD, Principal Investigator — Hospital de Niños Ricardo Gutierrez
Locations (3):
- Argentina (3):
  - Clinica y maternidad Suizo Argentina, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Materno Infantil Ramón Sardá, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital de Niños Ricardo Gutiérrez, Ciudad Autonoma de Buenos Aires, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salmerón MB. Estimación de prevalencia de infección congénita por citomegalovirus y seroprevalencia materna en Tucumán. Rev Argent Salud Pública. 2021;13:e33.
- [Background] Marín y col. - Citomegalovirosis congénita en población asintomática de recién nacidos de un hospital público en la Región Nordeste de Argentina. Rev Argent salud Pública, 2014; 5(20): 6-10
- [Result] Manicklal S, Emery VC, Lazzarotto T, Boppana SB, Gupta RK. The "silent" global burden of congenital cytomegalovirus. Clin Microbiol Rev. 2013 Jan;26(1):86-102. doi: 10.1128/CMR.00062-12. PMID 23297260
- [Result] Kenneson A, Cannon MJ. Review and meta-analysis of the epidemiology of congenital cytomegalovirus (CMV) infection. Rev Med Virol. 2007 Jul-Aug;17(4):253-76. doi: 10.1002/rmv.535. PMID 17579921
- [Result] Stagno S, Pass RF, Dworsky ME, Henderson RE, Moore EG, Walton PD, Alford CA. Congenital cytomegalovirus infection: The relative importance of primary and recurrent maternal infection. N Engl J Med. 1982 Apr 22;306(16):945-9. doi: 10.1056/NEJM198204223061601. PMID 6278309
- [Result] Wang C, Zhang X, Bialek S, Cannon MJ. Attribution of congenital cytomegalovirus infection to primary versus non-primary maternal infection. Clin Infect Dis. 2011 Jan 15;52(2):e11-3. doi: 10.1093/cid/ciq085. PMID 21288834
- [Result] Rawlinson WD, Boppana SB, Fowler KB, Kimberlin DW, Lazzarotto T, Alain S, Daly K, Doutre S, Gibson L, Giles ML, Greenlee J, Hamilton ST, Harrison GJ, Hui L, Jones CA, Palasanthiran P, Schleiss MR, Shand AW, van Zuylen WJ. Congenital cytomegalovirus infection in pregnancy and the neonate: consensus recommendations for prevention, diagnosis, and therapy. Lancet Infect Dis. 2017 Jun;17(6):e177-e188. doi: 10.1016/S1473-3099(17)30143-3. Epub 2017 Mar 11. PMID 28291720
- [Result] Boppana SB, Ross SA, Fowler KB. Congenital cytomegalovirus infection: clinical outcome. Clin Infect Dis. 2013 Dec;57 Suppl 4(Suppl 4):S178-81. doi: 10.1093/cid/cit629. PMID 24257422
- [Result] Fowler KB, McCollister FP, Dahle AJ, Boppana S, Britt WJ, Pass RF. Progressive and fluctuating sensorineural hearing loss in children with asymptomatic congenital cytomegalovirus infection. J Pediatr. 1997 Apr;130(4):624-30. doi: 10.1016/s0022-3476(97)70248-8. PMID 9108862
- [Result] Cannon MJ, Schmid DS, Hyde TB. Review of cytomegalovirus seroprevalence and demographic characteristics associated with infection. Rev Med Virol. 2010 Jul;20(4):202-13. doi: 10.1002/rmv.655. PMID 20564615
- [Result] Gantt S, Dionne F, Kozak FK, Goshen O, Goldfarb DM, Park AH, Boppana SB, Fowler K. Cost-effectiveness of Universal and Targeted Newborn Screening for Congenital Cytomegalovirus Infection. JAMA Pediatr. 2016 Dec 1;170(12):1173-1180. doi: 10.1001/jamapediatrics.2016.2016. PMID 27723885
- [Result] Boppana SB, Ross SA, Shimamura M, Palmer AL, Ahmed A, Michaels MG, Sanchez PJ, Bernstein DI, Tolan RW Jr, Novak Z, Chowdhury N, Britt WJ, Fowler KB; National Institute on Deafness and Other Communication Disorders CHIMES Study. Saliva polymerase-chain-reaction assay for cytomegalovirus screening in newborns. N Engl J Med. 2011 Jun 2;364(22):2111-8. doi: 10.1056/NEJMoa1006561. PMID 21631323
- [Result] Pinninti SG, Ross SA, Shimamura M, Novak Z, Palmer AL, Ahmed A, Tolan RW Jr, Bernstein DI, Michaels MG, Sanchez PJ, Fowler KB, Boppana SB; National Institute on Deafness and Other Communication Disorders CMV and Hearing Multicenter Screening (CHIMES) Study. Comparison of saliva PCR assay versus rapid culture for detection of congenital cytomegalovirus infection. Pediatr Infect Dis J. 2015 May;34(5):536-7. doi: 10.1097/INF.0000000000000609. PMID 25876092
- [Result] Ross SA, Ahmed A, Palmer AL, Michaels MG, Sanchez PJ, Bernstein DI, Tolan RW Jr, Novak Z, Chowdhury N, Fowler KB, Boppana SB; National Institute on Deafness and Other Communication Disorders CHIMES Study. Detection of congenital cytomegalovirus infection by real-time polymerase chain reaction analysis of saliva or urine specimens. J Infect Dis. 2014 Nov 1;210(9):1415-8. doi: 10.1093/infdis/jiu263. Epub 2014 May 5. PMID 24799600
- [Result] Yamamoto AY, Mussi-Pinhata MM, Marin LJ, Brito RM, Oliveira PF, Coelho TB. Is saliva as reliable as urine for detection of cytomegalovirus DNA for neonatal screening of congenital CMV infection? J Clin Virol. 2006 Jul;36(3):228-30. doi: 10.1016/j.jcv.2006.03.011. Epub 2006 Jun 5. PMID 16750653
- [Result] Belec L, Brogan TV. Real-time PCR-based testing of saliva for cytomegalovirus at birth. Expert Rev Anti Infect Ther. 2011 Dec;9(12):1119-24. doi: 10.1586/eri.11.130. PMID 22114962
- [Result] Barbi M, Binda S, Primache V, Caroppo S, Dido P, Guidotti P, Corbetta C, Melotti D. Cytomegalovirus DNA detection in Guthrie cards: a powerful tool for diagnosing congenital infection. J Clin Virol. 2000 Sep 1;17(3):159-65. doi: 10.1016/s1386-6532(00)00089-5. PMID 10996112
- [Result] Boppana SB, Ross SA, Novak Z, Shimamura M, Tolan RW Jr, Palmer AL, Ahmed A, Michaels MG, Sanchez PJ, Bernstein DI, Britt WJ, Fowler KB; National Institute on Deafness and Other Communication Disorders CMV and Hearing Multicenter Screening (CHIMES) Study. Dried blood spot real-time polymerase chain reaction assays to screen newborns for congenital cytomegalovirus infection. JAMA. 2010 Apr 14;303(14):1375-82. doi: 10.1001/jama.2010.423. PMID 20388893